CLINICAL TRIAL: NCT00549016
Title: Clinical Study of Aneurysm Exclusion Using PTFE Encapsulation of Nitinol Stents
Brief Title: Clinical Study of Aneurysm Exclusion
Acronym: EndoMed
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Arizona Heart Institute (Other)
Responsible Party: Edward B. Diethrich, MD, Arizona Heart Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G020035
Record Dates: First submitted 2007-10-24; First posted 2007-10-25 (Estimated); Last update posted 2009-05-15 (Estimated); Status verified 2009-05

CONDITIONS: Aneurysm
Keywords: Aneurysm Exclusion
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Device: PTPE Encapsulation of Nitinol Stents

INTERVENTIONS:
Device: PTPE Encapsulation of Nitinol Stents — Both common femoral arteries (CFAs) are surgically exposed to allow bilateral access of diagnostic and therapeutic devices. The endoluminal stent graft is then deployed in accordance with the Instructions for Use.

SUMMARY:
The ultimate purpose is to explore the potential techniques to exclude aneurysms and provide an alternative conduit for arterial flow. The single center sponsorship is intended to provide the investigators the potential to incorporate improvements in existing technology during the course of the study thereby ultimately enhancing the potential for superior medical care of patients suffering from these disease states. The sponsor/investigator recognizes and accepts responsibility to notify and receive approval from the agency when device modifications are made that may affect patient safety.

DETAILED DESCRIPTION:
The Arizona Heart Institute is respectfully submitting this protocol for a feasibility study utilizing the endoluminal grafts constructed of PTFE encapsulated nitinol stents. The study is intended to evaluate the use of this unique device in the treatment of aortic aneurysmal disease. The stent graft is made by laminating a PTFE "jacket" around nitinol stents which act as structural and fixation supports. Both materials have an extensive history of use in various types of implanted devices. CT scans and angiography or 3D computer imaging, and possibly IVUS imaging will be used to choose the sites for placement of the devices and to assure precise deployment.

In comparison to the conventional surgical approach, endoluminal stent-graft techniques for repair of abdominal aortic aneurysms (AAAs) offer the advantages of a minimally invasive procedure with lower morbidity and perhaps cost reduction. The Arizona Heart Institute has a long history in the area of endoluminal grafting for treatment of aneurysms and occlusive disease. Endoluminal sleeves principally using ePTFE and both stainless steel and nitinol stent structures have been studied using commercially available materials customized for particular pathologic situations. As the technology advances however, sophisticated engineering beyond the capabilities of our institution was required.

The proposed project originates because of the potential to escalate the combination of ePTFE and stents to a higher level of performance in aneurysm exclusion procedures. Current data reflect several deficiencies in approved exclusion devices. Migration, types I, II and III endoleaks and continual aneurysm expansion are clear predictors for potential ruptures. Increased complications associated with the initial peri-procedural deployment as devices are released on a broader scale have been observed. In order to address these problems, the Arizona Heart Institute has engaged EndoMed engineering to design the endoluminal graft to repair abdominal aortic aneurysms. We believe this will result in a positive step forward in the technology to exclude aneurysmal disease less invasively.

The endoluminal stent-graft is composed of multiple nitinol stents which are encapsulated in expanded Polytetrafluoroethylene (ePTFE). The stents are composed of a Z-shaped, performed nitinol wire, which is crimped together with a stainless steel sleeve to form the circular frame of the graft. This frame is then encapsulated between two thin sheets of laminated PTFE. The proximal end of the endoluminal stent-graft is made in two configurations. One is a completely encapsulated graft where the PTFE covers the entire device. The other has an open stent segment (bare wire configuration) that allows the open stent region of the graft to be placed across the orifice of the renal, mesenteric, or internal iliac arteries without obstructing antegrade blood flow. The device will be available in a straight tube, aortomonoiliac or bifurcated design.

Once the endoluminal stent graft is built, a 4 French guidewire dilator is placed through the center of the graft and the assembly is compressed into a high density polyethylene (HDPE) cartridge for ease of intraluminal delivery. The endoluminal stent-graft is then placed in two Tyvek pouches and sterilized using Hydrogen Peroxide.

Subjects will undergo an evaluation of the PTFE encapsulation of Nitinol stents to provide data on the device's feasibility for therapeutic clinical use. Follow-up will be completed at 1, 6, 12, 24, 36, 48, and 60 months. Subject evaluation at 1 month will include a Complete History and Physical, Bilateral ABIs, Abdominal Duplex Ultrasound, and a KUB X-ray (4 views). Subject evaluation at 6 months will also include a Complete History and Physical, Bilateral ABIs, Abdominal Duplex Ultrasound, KUB X-ray (4 views), and based on the duplex ultrasound an Abdominal CT scan with and without IV contrast 2.5 mm and Labs (BUN/Creatinine). Subject evaluation at 12, 24, 36, 48, and 60 months will include a Complete History and Physical, Bilateral ABIs, Abdominal CT scan with and without IV contrast 2.5 mm, Abdominal Duplex Ultrasound, KUB X-ray (4 views), and Labs (BUN/Creatinine).

ELIGIBILITY:
Inclusion Criteria:

* Aneurysm diameter ≥ 4.0 cm; or aneurysm diameter ≤ 4.0 cm which has exhibited rapid expansion; or aneurysms with saccular configuration where potential for rupture is increased; or aneurysms which have exhibited dissection and there is potential for rupture or compromised flow to vital structures; or symptomatic leaking or ruptured aneurysms.
* Vessels proximal and distal to the lesion must be capable of accommodating the device.
* The access artery diameter and profile of the artery must be capable of the device delivery.
* Patients must be ASA III or higher.
* Informed consent must be obtainable.
* Patients must be willing and able to comply with the follow-up regime.
* Patients with neck grades as follow:
* Grade I: Length of Proximal Neck ≥ 1.5 cm and Distal Neck ≥ 1.0 cm
* Grade II: Length of Proximal Neck ≥ 1.5 cm, but Distal Neck < 1.0 cm without obvious iliac aneurysms, or aneurysm extends into or is associated with iliac aneurysms.
* Grade III: Length of Proximal Neck < 1.5 cm and Distal Neck ≥ 1.0 cm
* Grade IV: Length of Proximal Neck < 1.5 cm and Distal Neck < 1.0 cm or the involvement as in Grade II.

Exclusion Criteria:

* A proximal neck less than 0.5 cm in length.
* Arterial diameter larger than 40 mm at the proximal or distal landing zones.
* Iliac diameter less than 6 mm (following balloon angioplasty as needed).
* The inferior mesenteric artery is indispensable.
* Patients under the age of 18.
* Pregnant or lactating women.
* Patients with allergy to any of the device materials.
* Patients with uncorrectable coagulopathy or bleeding disorders.
* Patients for whom contrast medium or anticoagulation drugs are contraindicated.
* Patients with active systemic or localized groin infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2002-11; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Technical success in the deployment and placement of the endoluminal graft to the aneurysmal site. | 1 month

SECONDARY OUTCOMES:
Acute success when the endoluminal graft excludes the aneurysm and maintain patency without endoleaks, migration or rupture. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Edward B Diethrich, M.D., Principal Investigator — Arizona Heart Institute
Locations (1):
- Arizona Heart Institute, Phoenix, Arizona, United States